CLINICAL TRIAL: NCT03620604
Title: Mid Term Safety and Efficacy of ALTIS® Single Incision Sling for Female SUI. Less Mesh, Same Results.
Brief Title: Mid Term Safety and Efficacy of ALTIS® Single Incision Sling for Female Stress Urinary Incontinence (SUI).
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Principal Investigator, Eduardo Moran, Urologist, Instituto de Investigacion Sanitaria La Fe
Other Study IDs: ALTIS STUDY
Record Dates: First submitted 2018-07-28; First posted 2018-08-08 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Urinary Incontinence,Stress
Keywords: single incision sling; safety; efficacy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Stress urinary incontinence surgery: This is a single observational study were all patients had stress urinary incontinence. All of them underwent surgery performing a single incision sling type ALTIS
  Interventions: Device: Stress urinary incontinence surgery

INTERVENTIONS:
Device: Stress urinary incontinence surgery — All patients were treated according to the Urology protocols of our unit. They were patients with stress urinary incontinence refractory to pelvic floor exercises so they underwent surgery
  Other Names: ALTIS device

SUMMARY:
Prospective, single-arm, non-sponsored, observational single centre trial in a cohort of patients undergoing stress urinary incontinence surgery with ALTIS® procedure. All patients were diagnosed according to clinical reports, physical exploration and urodynamics. Body mass index(BMI) was categorized according to World Health Organization classification. Valsalva leak point pressure was categorized in three groups <60 cmH2O, 60-90 cmH2O and >90 cmH2O). Participants were evaluated post-operatively at 1, 6, 12 and 24 months with physical examination, ICIQ-SF, visual scale of satisfaction(SVS)(0-10). Adverse events were reported in each visit. Multivariate analysis for risk factors of surgery failure was performed.

DETAILED DESCRIPTION:
This is a prospective, single -arm, non-sponsored observational single centre trial in a cohort of patients undergoing stress urinary incontinence surgery with ALTIS® procedure. Two urologists, experts in female incontinence surgery, performed all procedures. Safety and efficacy were evaluated. All participants provided written informed consent prior to enrolment.

The investigators recruited female patients aged 35 years or more with urodynamically proven stress urinary incontinence and who had failed to 6 months of non-surgical therapies including behavioural changes and drug therapy. Exclusion criteria were pelvic infection, pelvic organ prolapse ≥Stage 2, prior stress urinary incontinence surgery, neurogenic bladder incontinence, previous pelvic radiotherapy, high post-voiding volume (100 mL in two times) or being pregnant.

Demographic variables (age, number of vaginal deliveries, prior stress urinary incontinence surgery, menopause status, BMI and presence of urge incontinence) were collected. BMI was categorized according to World Health Organization in normal (18,5-24,9 Kg/m2), overweight (25-29,9 Kg/m2) and obese (≥ 30 Kg/m2) patients. For statistical purpose the investigators divided patients into two groups, non-obese (18,5-29,9) Kg/m2) and obese (≥ 30 Kg/m2) patients.

Preoperative assessment included urogynecological history, cough test (stress test with at least 300 mL of bladder volume measured by ultrasound), Spanish validated version of the International Consultation on Incontinence Questionnaire sort form (ICIQ-SF) and urodynamic test (Urodynamic parameters as Valsalva leak point pressure (VLPP), non-inhibited detrusor contractions and post-voiding volume were reflected. VLPP was categorized into three groups <60 cmH2O, 60-90 cmH2O and >90 cmH2O).

Follow up was carried out with physical examination, ICIQ-SF, visual scale of satisfaction and physical examination including cough test. Subjects were evaluated post-operatively at 1, 6, 12 and 24 months. Adverse events, such as vaginal erosion or pain related to the procedure or the device were evaluated at each visit.

The primary efficacy measures were objective cure, defined as negative cough test, and subjective cure, defined as ICIQ-SF=0.

ELIGIBILITY:
Inclusion Criteria:

* Urodynamically proven stress urinary incontinence
* Refractory to 6 months of non-surgical therapies including behavioural changes or drug therapy

Exclusion Criteria:

* Pelvic infection
* Pelvic organ prolapse ≥Stage 2
* Prior stress urinary incontinence surgery
* Neurogenic bladder incontinence,
* Previous pelvic radiotherapy,
* High post-voiding volume (100 mL in two times)
* Pregnant women.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were selected from our National Health System both forwarded from primary care or f from gynecology or other urologist to de Urodynamic Unit
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mid term Efficacy/continence | Assessed at 24 months of follow up
  Mid term Efficacy and continence measured with cough test ( Positive or negative)

SECONDARY OUTCOMES:
Voiding disfunction | Assessed every visit at 1,6,12,24 months
  Difficulty to void assessed by uroflowmetry (mL/s)
De novo urgency | Assessed at visit 6,12,24 months
  measured by International Consultation on Incontinence Questionnaire Sort Form (ICIQ-SF) ( from 0 to 21 being 0 = to continence and 21= the worse outcome of incontinence)
Safety and adverse events | Assessed every visit at 1,6,12,24 months
  Safety was assessed by physical examination to rule out vaginal extrusion (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo J Moran Pascual, Doctor, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Hospital Universitario y Politecnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
This is a single centre study we don't think it will be useful to make these data available to other researchers

REFERENCES:
- [Background] Kocjancic E, Erickson T, Tu LM, Gheiler E, Van Drie D. Two-year outcomes for the Altis(R) adjustable single incision sling system for treatment of stress urinary incontinence. Neurourol Urodyn. 2017 Aug;36(6):1582-1587. doi: 10.1002/nau.23156. Epub 2016 Oct 29. PMID 27794177
- [Background] Van Drie DM. The Impact of Procedure Setting on Two-Year Outcomes for the Altis Single Incision Sling for Women With Stress Urinary Incontinence. J Minim Invasive Gynecol. 2015 Nov-Dec;22(6S):S243-S244. doi: 10.1016/j.jmig.2015.08.853. Epub 2015 Oct 15. No abstract available. PMID 27679164
- [Background] Dias J, Xambre L, Costa L, Costa P, Ferraz L. Short-term outcomes of Altis single-incision sling procedure for stress urinary incontinence: a prospective single-center study. Int Urogynecol J. 2014 Aug;25(8):1089-95. doi: 10.1007/s00192-014-2355-4. Epub 2014 Mar 6. PMID 24599178